CLINICAL TRIAL: NCT02812381
Title: Efficacy of Neuromuscular Bandage Technique Against Jones Technique After the Supraespinatus Muscle Tendon Suture: a Prospective Randomized Clinical Trial
Brief Title: Efficacy of Neuromuscular Bandage Technique Against Jones Technique After the Supraespinatus Muscle Tendon Suture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC-2013
Record Dates: First submitted 2016-03-29; First posted 2016-06-24 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-03

CONDITIONS: Pain
Keywords: Trigger Points, movement
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCS (Jones tecnique) (Active Comparator): 18 patients were treatment with straincounterstrain
  Interventions: Procedure: SCS
- KT Kinesiotaping (Sham Comparator): 18 patients were treatment with neuromuscular bandage
  Interventions: Procedure: KT

INTERVENTIONS:
Procedure: KT — to aplicate neuromuscular bandage technique(KT)
  Arms: KT Kinesiotaping
Procedure: SCS — To aplicate strain-counterstrain above trigger point
  Arms: SCS (Jones tecnique)

SUMMARY:
The suture of the supraspinatus tendon is a common surgery that requires physical therapy for back pain and functional impairment to such surgery. Kinesiotaping technique (KT) is being used to treat myofascial trigger points that appear after surgery and for the treatment of physiotherapy in the supraspinatus muscle and deltoid.

To evaluate the effectiveness of KT technique over the technique of Jones (Straincounterstrain or SCS) in patients undergoing suture the tendon of the supraspinatus muscle.

DETAILED DESCRIPTION:
Objective: To evaluate the effectiveness of the KT technique against Jones (Strain-Counterstrain or SCS) technique in patients with the suture of the tendon of the supraspinatus muscle.

Design: Test clinically controlled, randomized, masking of intervention by double placebo and blind to the subject of the essay and the Studio analyst.

METHOD: Patients with supraspinatus tendon suture are randomly divided into two groups: a group treated with KT (n = 18) and other treated with SCS (n = 18). The treatment was applied the 1st, 4th and 8th day of physical therapy session. All patients were evaluated the 1st and the 12th day of the session with the visual analog scale of pain (VAS), with the scale of Disabilities of the arm, shoulder and hand (DASH) to assess the functionality and active direction-finding (ROM) to assess travel articulate.

ELIGIBILITY:
Inclusion Criteria:

* Among patients attending the 1st and 5th week after Intervention.
* Patients with age above 18 years.
* Patients of both sexes.
* Patients with a detectable with algometer trigger point in the supraspinatus and / or deltoid .

Exclusion Criteria:

* Patient with Impaired Communication .
* Patients with signs of infection .
* Patients with previous surgery on the shoulder or shoulder capsulitis submit .
* Patient scammers cervical herniated discs or brachial neuropathy .
* Patients with tumor pathology.
* Patients with fibromyalgia,
* Pregnant patients.
* Patients with central pain .
* Patients conducted simultaneously treatments .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in the DASH between sixth and eighth week , in patients with supraespinatus muscle tendon suture. | From first day of the sixth week after surgery to twelve days after of the first medition.
  All participants (36) has been mesured:
  * First day of the sixth week after surgery with DASH,
  * Four days later of the first medition , it repeated the technique asigned but it hasn´t been mesured.
  * Eight days later or the first meditión, it repeated the technique asigned but it hasn´t been mesured.
  * Twelve days later of the first medition , it repeated the mesured with DASH,

SECONDARY OUTCOMES:
Change in the VAS between sixth and eighth week , in patients with supraespinatus muscle tendon suture. | From first day of the sixth week after surgery to twelve days after of the first medition.
  All participants (36) has been mesured:
  * First day of the sixth week after surgery with VAS scale.
  * Four days later of the first medition , it repeated the technique asigned but it hasn´t been mesured.
  * Eight days later or the first meditión, it repeated the technique asigned but it hasn´t been mesured.
  * Twelve days later of the first medition , it repeated the mesured with VAS

OTHER OUTCOMES:
Change in the ROM between sixth and eighth week , in patients with supraespinatus muscle tendon suture. | From first day of the sixth week after surgery to twelve days after of the first medition.
  All participants (36) has been mesured:
  * First day of the sixth week after surgery with ROM
  * Four days later of the first medition , it repeated the technique asigned but it hasn´t been mesured.
  * Eight days later or the first meditión, it repeated the technique asigned but it hasn´t been mesured.
  * Twelve days later of the first medition , it repeated the mesured with ROM

CONTACTS AND LOCATIONS:
Overall Officials: ANA ROMOJARO, THERAPIST, Principal Investigator — UNIVERSIDAD DE ALCALA

IPD SHARING:
Plan to Share IPD: Yes
The investigators would like to share in the magazine "Manual Therapy"